CLINICAL TRIAL: NCT03843125
Title: A Phase 3, Double-Blind, Multicenter Study to Evaluate the Long-Term Safety and Efficacy of Baricitinib in Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: A Study of Baricitinib in Participants With Systemic Lupus Erythematosus (SLE)
Acronym: SLE-BRAVE-X
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to insufficient evidence to support a positive benefit: risk profile. Safety findings were consistent with previously published OLUMIANT data
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16832; I4V-MC-JAIM (Other: Eli Lilly and Company); 2017-005028-11 (EudraCT Number)
Record Dates: First submitted 2019-02-14; First posted 2019-02-15 (Actual); Results first posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 2 mg Baricitinib (Experimental): Participants received one 2 mg Baricitinib tablet and one placebo tablet matching 4 mg Baricitinib administered orally every day (QD).
  Interventions: Drug: Baricitinib; Drug: Placebo
- 4 mg Baricitinib (Experimental): Participants received one 4 mg Baricitinib tablet and one placebo tablet matching 2 mg Baricitinib administered orally QD.
  Interventions: Drug: Baricitinib; Drug: Placebo
- Placebo to 2 mg Baricitinib (Experimental): Participants who received placebo in the originating study (JAHZ or JAIA) were randomized to receive 2 mg Baricitinib administered orally QD.
  Interventions: Drug: Baricitinib; Drug: Placebo
- Placebo to 4 mg Baricitinib (Experimental): Participants who received placebo in the originating study (JAHZ or JAIA) were randomized to receive 4 mg Baricitinib administered orally QD.
  Interventions: Drug: Baricitinib; Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Administered orally.
  Other Names: LY3009104
Drug: Placebo — Administered orally.

SUMMARY:
The reason for this long term study is to see how safe and effective the study drug known as baricitinib is in participants with systemic lupus erythematosus (SLE) who have completed the final treatment visit of study I4V-MC-JAHZ (NCT03616912) or study I4V-MC-JAIA (NCT03616964).

ELIGIBILITY:
Inclusion Criteria:

* Have completed the final treatment study visit of an originating study, such as study JAHZ (NCT03616912) or Study JAIA (NCT03616964).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1147 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (297):
- United States (61):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Arizona Arthritis & Rheumatology Research, Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Associates, P. C., Tucson, Arizona
  - Wallace Rheumatic Studies Center, Beverly Hills, California
  - Medvin Clinical Research - Weidmann, Covina, California
  - Providence Medical Foundation, Fullerton, California
  - MD Medical Corporation, Hemet, California
  - ACRC Studies, Poway, California
  - Inland Rheumatology & Osteoporosis Medical Group, Upland, California
  - Medvin Clinical Research - Weidmann, Whittier, California
  - Denver Arthritis Clinic - Lowry, Denver, Colorado
  - New England Research Associates, Bridgeport, Connecticut
  - Arthritis and Rheumatic Disease, Aventura, Florida
  - Clinical Research of West Florida, Inc. (Clearwater), Clearwater, Florida
  - Lakes Research, LLC, Miami Lakes, Florida
  - Millennium Research, Ormond Beach, Florida
  - Integral Rheumatology & Immunology Specialists, Plantation, Florida
  - IRIS Research and Development, LLC, Plantation, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Tampa Medical Group, P.A., Tampa, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - North Georgia Rheumatology, PC, Lawrenceville, Georgia
  - Arthritis Center of Lexington, Lexington, Kentucky
  - Johns Hopkins Asthma and Allergy Center, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Advanced Rheumatology, PC, Lansing, Michigan
  - Clinical Research Institute of Michigan, LLC, Saint Clair Shores, Michigan
  - Glacir View Research Institute, Kalispell, Montana
  - Allied Clinical Research, Reno, Nevada
  - Arthritis and Osteoporosis Associates of New Mexico, Las Cruces, New Mexico
  - St. Lawrence Health System, Canton, New York
  - The Feinstein Institute for Medical Research, Manhasset, New York
  - Columbia University Medical Center, New York, New York
  - NYU Langone, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Joint and Muscle Medical Care, Charlotte, North Carolina
  - Box Arthritis & Rheumatology of the Carolinas, PLLC, Charlotte, North Carolina
  - Medication Management, Greensboro, North Carolina
  - Cincinnati Rheumatic Disease Study Group, Cincinnati, Ohio
  - Paramount Medical Research, Middleburg Heights, Ohio
  - Arthritis & Rheumatology Center of Oklahoma PLLC, Oklahoma City, Oklahoma
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - East Penn Rheumatology Associates, Bethlehem, Pennsylvania
  - Clinical Research Center of Reading,LLC, Wyomissing, Pennsylvania
  - Articularis Healthcare d/b/a/ Low Country Rheumatology, PA, Summerville, South Carolina
  - Eagle Medical, Crossville, Tennessee
  - West Tennessee Research Institute, Jackson, Tennessee
  - Amarillo Center for Clinical Research, Amarillo, Texas
  - Accurate Clinical Management, Baytown, Texas
  - Dr. Dhiman Basu Private Practice, Colleyville, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Precision Comprehensive Clinical Research Solutions, Fort Worth, Texas
  - Rheumatology Center Of Houston, Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Southwest Rheumatology, P.A., Mesquite, Texas
  - Accurate Clinical Research, Inc., San Antonio, Texas
  - Advanced Rheumatology of Houston, The Woodlands, Texas
  - Arthritis Clinic of Northern VA, P.C., Arlington, Virginia
  - Spectrum Medical Inc., Danville, Virginia
  - Rheumatic Disease Center, Glendale, Wisconsin
- Argentina (10):
  - Aprillus Asistencia e Investigacion de Arcis Salud SRL, Ciudad Autónoma de Buenos Aire, Buenos Aires
  - DOM Centro de Reumatologia, Ciudad de Buenos Aires, Buenos Aires
  - Framingham Centro Medico, La Plata, Buenos Aires
  - CER Instituto Medico, Quilmes, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes, Buenos Aires
  - Clinica Adventista Belgrano, CABA, Ciudad Autónoma de Buenos Aire
  - Sanatorio Británico, Rosario, Santa Fe Province
  - Centro de Educación Médica e Investigaciones Clínicas "Norberto Quirno" (CEMIC), Buenos Aires
  - IR Medical Center S.A. Instituto de Reumatologia, Mendoza
  - Centro de Investigaciones Médicas Tucuman, San Miguel de Tucumán
- Australia (4):
  - Optimus Clinical Research, Botany, New South Wales
  - The Rheumatology Research Unit Sunshine Coast, Maroochydore, Queensland
  - Emeritus Research, Camberwell, Victoria
  - St. Vincent's Hospital, Fitzroy, Victoria
- Austria (2):
  - A O Krankenhaus der Elisabethinen, Linz, Upper Austria
  - Medizinische Universität Graz, Graz
- Belgium (2):
  - UZ Leuven, Leuven, Vlaams Brabant
  - Cliniques Universitaires Saint-Luc, Brussels
- Brazil (7):
  - SER - Serviços Especializados em Reumatologia da Bahia S/S - ME, Salvador, Estado de Bahia
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Centro de Estudos em Terapias Inovadoras-CETI, Curitiba, Paraná
  - EDUMED - Educação em Saúde Ltda., Curitiba, Paraná
  - LMK Serviços Médicos S/S, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas UNICAMP, Campinas, São Paulo
  - Oncovida- Centro de Onco-Hematologia de Mato Grosso, Cuiabá
- Chile (6):
  - Clinical Research Chile SpA, Valdivia, Los Ríos Region
  - Enroll SpA, Providencia, Región Metropolitana de Santia
  - Clinica Alemana de Osorno, Osorno
  - Sociedad Medica Del Aparato Locomotor SA, Santiago
  - Prosalud y cia. Ltda., Santiago
  - CINVEC- Estudos Clínicos Quinta Región Limitada, Viña del Mar
- China (17):
  - The First Affliated Hospital of Suzhou University, Suzhou, China
  - First affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - First Affiliated Hospital of the Harbin Medical University, Harbin, Heilongjiang
  - Wuhan Union Hospital, Wuhan, Hubei
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - China-Japan Union Hospital, CJUH., Changchun, Jilin
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Peking University First Hospital, Beijing
  - Beijing Peking Union Medical College Hospital, Beijing
  - Shanghai Huashan Hospital Affil to Fu Dan University, Shanghai
  - China Medical University (CMU) - First Affiliated Hospital, Shenyang
  - The First Affiliated Hospital of Zhengzhou Universtiy, Zhengzhou
- Colombia (7):
  - HPTU-El Hospital con alma Pablo Tobon Uribe, Medellín, Antioquia
  - Clinica de la Costa, Barranquilla, Atlántico
  - Circaribe SAS, Barranquilla, Atlántico
  - Idearg S.A.S., Bogota, Cundinamarca
  - Servimed S.A.S., Bucaramanga, Santander Department
  - Centro de Medicina Interna, Cali, Valle del Cauca Department
  - Preventive Care Ltdac, Chía
- Croatia (2):
  - Klinicki Bolnicki Centar Rijeka, Rijeka
  - University Hospital Split, Split
- Czechia (5):
  - Revmatologicky ustav, Prague, Praha, Hlavní Mešto
  - Revmatologie.s.r.o., Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - ARTHROHELP s.r.o., Pardubice
  - VFN a 1 LF University Karlovy, Prague
- France (5):
  - CHRU Brest - Hopital Cavale Blanche, Brest, Finistère
  - Centre hospitalier universitaire Pellegrin, Bordeaux
  - CHRU Lille - Hopital Claude Huriez, Lille
  - Hopital Européen, Marseille
  - Hôpital de HautePierre, Strasbourg
- Germany (11):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Klinikum der Universität München Großhadern, München, Bavaria
  - Universitätsklinikum Würzburg A. ö. R., Würzburg, Bavaria
  - Universitätsmedizin Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universitatsklinikum Leipzig, Leipzig, Saxony
  - Charité Campus Virchow-Klinikum, Berlin
  - Immanuel Krankenhaus Rheuma Klinik Berlin Buch, Berlin
  - Schlosspark Klinik, Berlin
  - Universitaetsklinikum Koeln, Cologne
- Greece (5):
  - Gen Hospital of Athens G Gennimatas, Athens, Attica
  - University General Hospital of Heraklion, Heraklion, Irakleío
  - Regional General University Hospital of Larissa, Larissa
  - Kianous Stavros, Thessaloniki
  - Gen. Hosp. of Thessaloniki "Hippokration", Thessaloniki
- Hungary (10):
  - Békés Megyei Központi Kórház Pándy Kálmán Tagkórház, Gyula, Bekes County
  - Vital Medical Center, Veszprém, Veszprém City
  - Budai Irgalmasrendi Korhaz, Budapest
  - Qualiclinic, Budapest
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Budapest
  - Debreceni Egyetem Orvos-es Egészsegtudomanyi Centrum, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont I. Belgyogyaszati Klinika, Szeged
  - Vita Verum Egeszsegugyi Szolgaltato Bt, Székesfehérvár
- India (13):
  - Panchshil hospital, Ahmedabad, Gujarat
  - CIMS Hospital Private Limited, Ahmedabad, Gujarat
  - Shree Giriraj Hospital, Rajkot, Gujarat
  - Nirmal Hospital Private Limited, Surat, Gujarat
  - Sterling Hospital, Vadodara, Gujarat
  - ChanRe Rheumatology And Immunology Center And Research, Bangalore, Karnataka
  - St. John Medical College & Hospital, Bangalore, Karnataka
  - Sushruta Multispecialty Hospital & Research Center Pvt Ltd, Hubli, Karnataka
  - Kasturba Medical College Hospital, Mangalore, Madhav Nagar, Manipal, Karnataka
  - Jasleen Hospital, Nagpur, Maharashtra
  - Synexus Affiliate - Sujata Birla Hospital & Medical Research Center, Nashik, Maharashtra
  - Fortis Escorts Hospital, Jaipur, Rajasthan
  - Krishna Institute of Medical Science, Secunderabad, Telangana
- Israel (3):
  - Meir Medical Center, Kfar Saba
  - Sheba Medical Center, Ramat Gan
  - Carmel Hospital, Haifa, Ḥeifā
- Italy (4):
  - Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Azienda Policlinico Umberto I, Roma
  - Azienda Ospedaliera Santa Maria Della Misericordia, Udine
- Japan (17):
  - University of Occupational and Enviromental Health, Kitakyushu, Fukuoka
  - National Hospital Organization Asahikawa Medical Center, Asahikawa, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Jp Red Cross Society Himeji Hp, Himeji, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Tomishiro Central Hospital, Tomigusuku, Okinawa
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Nippon Medical School Hospital, Bunkyo-Ku, Tokyo
  - Showa University Hospital, Shinagawa, Tokyo
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Hamanomachi Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - St. Luke's International Hospital, Tokyo
  - Keio university hospital, Tokyo
- Mexico (16):
  - Dr. Alberto Esteban Bazzoni Ruiz, Torreón, Coahuila
  - Morales Vargas Centro de Investigacion, S.C., León, Guanajuato
  - Centro Integral en Reumatologia SA de CV, Guadalajara, Jalisco
  - Clinica de Investigacion en Reumatologia y Obesidad S. C., Guadalajara, Jalisco
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, Guadalajara, Jalisco
  - Investigación Biomédica para el Desarrollo de Fármacos S.A. de C.V., Zapopan, Jalisco
  - Clinica para el Diagnostico y Tratamiento de la Enfermedades, Mexico City, Mexico City
  - Centro de Alta Especialidad Reumatologia Inv del Potosi SC, San Luis Potosí City, San Luis Potosí
  - Consultorio Jose Luis Garcia Figueroa, Villahermosa, Tabasco
  - Centro Peninsular de Investigacion S.C.P, Mérida, Yucatán
  - Köhler & Milstein Research, Mérida, Yucatán
  - Cemdeicy S.C.P., Mérida, Yucatán
  - Clinosar Mexico S.A. de C.V, Mexico City
  - Consultorio de Reumatologia, Mexico City
  - Centro de Investigación y Tratamiento Reumatológico S.C, Mexico City
  - Oaxaca Site Management Organization, Oaxaca City
- Netherlands (2):
  - Medische Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - Vrije Universiteit Medisch Centrum Amsterdam, Amsterdam
- Philippines (7):
  - Mary Mediatrix Medical Center, Lipa, Batangas
  - Cebu Doctors Hospital, Cebu City, Cebu
  - Chong Hua Hospital, Cebu City, Cebu
  - Southern Philippines Medical Center, Davao City, Davao Del Norte
  - Makati Medical Center, Makati, Luzon
  - St. Luke's Medical Center, Quezon City, Luzon
  - Angeles University Foundation and Medical Center, Angeles City, Pampanga
- Poland (15):
  - Szpital Uniwersytecki Nr 2 im. dr J. Biziela w Bydgoszczy, Klinika Reumatologii i Chorob Tkanki Lacznej, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej Biogenes Sp. z o.o., Wroclaw, Lower Silesian Voivodeship
  - Twoja Przychodnia Centrum Medyczne Nowa Sol, Nowa Sól, Lubusz Voivodeship
  - Medycyna Kliniczna, Warsaw, Masovian Voivodeship
  - Reumatika - Centrum Reumatologii, Warsaw, Masovian Voivodeship
  - Gabinet Internistyczno- Reumatologiczny Piotr Adrian Klimiuk, Bialystok, Podlaskie Voivodeship
  - Zespol Poradni Specjalistycznych REUMED, Lublin, Polska
  - Ambulatorium Barbara Bazela, Elblag, Warminsko-Mazurki
  - Centrum Medyczne Pratia Katowice, Katowice
  - MCM Krakow - PRATIA - PPDS, Krakow
  - Centrum Medyczne Plejady, Krakow
  - NZOZ Lecznica MAK-MED s.c., Nadarzyn
  - Klinika Reumatologii i Rehabilitacji, Poznan
  - Klinika Reumatologii, Chorob Wewnetrznych i Geriatrii PUM, Szczecin
  - Centrum Medyczne AMED, Warsaw
- Romania (7):
  - C.M.D.T.A. Neomed, Brasov, Brașov County
  - Spitalul Euroclinic, Bucureti, București
  - Napoca Emergency Clinical County Hospital, Cluj-Napoca, Cluj
  - Craiova Emergency Clinical County Hospital, Craiova, Dolj
  - Spitalul Clinic Sf Maria Bucuresti, Bucharest
  - Spitalul Clinic "Dr. Ioan Cantacuzino", Bucharest
  - SANA Medical Center, Bucharest
- Russia (17):
  - Moscow City Clinical Hospital Number 52, Moscow, Moscow
  - Russian National Research Medical University n.a. N.I.Pirogov, Moscow, Russian Federation
  - LLC MK Med, Saint Petersburg, Sankt-Peterburg
  - Chelyabinsk Regional Clinical Hospital, Chelyabinsk
  - City Hospital # 7, Kazan'
  - V.A. Nasonova Research Institute of Rheumatology, Moscow
  - City Clinical Hospital 1 named after N.I. Pirogov, Moscow
  - Research Institute of Clinical Immunology, Novosibirsk
  - Institute of Cytology and Genetics of Siberian Branch of Russian Academy of Medical Sciences, Novosibirsk
  - Regional Hospital - Omsk, Omsk
  - Orenburg State Medical Academy of Roszdrav, Orenburg
  - Kursk Regional Clinical Hospital, Rursk
  - Ryazan State Medical University, Ryazan
  - Russian Medical Military Academy n.a. S.M. Kirov, Saint Petersburg
  - Departmental Hospital at Smolensk Station "rzhd" JSC, Smolensk
  - Kuvatov Republican Clinical Hospital, Ufa
  - LLC Medical Center Zdorovaya Semiya, Zonova
- Serbia (5):
  - Institute of Rheumatology, Belgrade
  - Military Medical Academy, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - Institute for Treatment and Rehabilitation Niska Banja, Niška Banja
  - Clinical Center of Vojvodina, Novi Sad
- South Africa (7):
  - Suite 509 Umhlanga Netcare Medical Centre, Umhlanga, Durban
  - WITS Clinical Research, Johannesburg, Gauteng
  - Jakaranda Hospital, Pretoria, Gauteng
  - Vincent Pallotti Hospital, Cape Town, Western Cape
  - Panorama Medical Centre, Cape Town, Western Cape
  - Winelands Medical Research Centre, Stellenbosch, Western Cape
  - University Of Pretoria, Pretoria
- South Korea (7):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Kyung Pook National University Hospital, Daegu, Korea
  - Chungnam National University Hospital, Daejeon, Korea
  - Gachon University Gil Hospital, Incheon, Korea
  - Hanyang University Medical Center, Seoul, Korea
  - Asan Medical Center, Seoul, Korea
  - Seoul St. Mary's Hospital, Seoul, Korea
- Spain (7):
  - Hospital Marina Baixa, Villajoyosa, Alicante
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Corporacion Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital De Fuenlabrada, Fuenlabrada, Madrid
  - Hospital do Meixoeiro, Vigo, Pontevedra
  - Corporació Sanitària Clínic, Barcelona
  - Hospital Quiron Infanta Luisa, Seville
- Cantonal Hospital St.Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland
- Taiwan (9):
  - Hualien Tzu-Chi Hospital, Dalin Township
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi-Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan
- United Kingdom (6):
  - Maidstone Hospital, Maidstone, Kent
  - Whipps Cross University Hospital, Leytonstone, London
  - St George's Hospital, Tooting, London
  - Guys/St. Thomas Hospital, London, Surrey
  - Doncaster and Bassetlaw Teaching Hospitals NHS Foundation Trust, Doncaster
  - Leeds Teaching Hospital, Leeds

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Baricitinib in Participants With Systemic Lupus Erythematosus (SLE) — https://trials.lillytrialguide.com/en-US/trial/522BW42nIOGg3wGqAYUcrw

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed originating study [I4V-MC-JAHZ (NCT03616912) or Study I4V-MC-JAIA (NCT03616964)] were enrolled in this study.
Pre-assignment Details: Participants who were randomized to placebo during originating Study I4V-MC-JAHZ (NCT03616912) or Study I4V-MC-JAIA (NCT03616964) were randomized 1:1 to receive baricitinib 4-milligrams (mg) or baricitinib 2-mg once daily (QD), administered orally.
Groups:
- 2 Milligrams (mg) Baricitinib: Participants received one 2 mg Baricitinib tablet and one placebo tablet matching 4 mg Baricitinib administered orally every day (QD).
Period: Overall Study
Arm/Group | 2 Milligrams (mg) Baricitinib | 4 mg Baricitinib | Placebo to 2 mg Baricitinib | Placebo to 4 mg Baricitinib
Started | 388 | 379 | 189 | 191
Safety Population (All participants who received at least one dose of study drug and who did not discontinue from the study for the reason 'Lost to Follow-up' at the first postbaseline visit.) | 388 | 378 | 189 | 191
Completed | 0 | 0 | 0 | 0
Not Completed | 388 | 379 | 189 | 191
Not completed — Adverse Event | 17 | 13 | 5 | 9
Not completed — Death | 0 | 6 | 2 | 0
Not completed — Lack of Efficacy | 14 | 11 | 9 | 4
Not completed — Lost to Follow-up | 3 | 4 | 0 | 2
Not completed — Other | 12 | 14 | 3 | 4
Not completed — Due to Epidemic/Pandemic | 1 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 318 | 318 | 163 | 163
Not completed — Withdrawal by Subject | 23 | 12 | 6 | 9
Not completed — Missing data | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 2 mg Baricitinib: Participants received one 2 mg Baricitinib tablet and one placebo tablet matching 4 mg Baricitinib administered orally QD.
- Total: Total of all reporting groups
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | Placebo to 2 mg Baricitinib | Placebo to 4 mg Baricitinib | Total
Number analyzed (Participants) | 388 | 379 | 189 | 191 | 1147
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (12.68) | 43.8 (12.03) | 43.8 (11.85) | 43.5 (13.22) | 43.7 (12.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 361 | 357 | 181 | 176 | 1075
  Male | 27 | 22 | 8 | 15 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 21 | 16 | 13 | 11 | 61
  Asian | 79 | 77 | 44 | 41 | 241
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 32 | 36 | 19 | 19 | 106
  White | 249 | 241 | 109 | 115 | 714
  More than one race | 3 | 2 | 2 | 2 | 9
  Unknown or Not Reported | 4 | 7 | 2 | 3 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 66 | 68 | 28 | 30 | 192
  Czechia | 7 | 9 | 7 | 5 | 28
  Russia | 19 | 16 | 11 | 11 | 57
  Greece | 8 | 4 | 0 | 3 | 15
  South Korea | 7 | 7 | 2 | 2 | 18
  Netherlands | 1 | 1 | 0 | 0 | 2
  Austria | 1 | 1 | 0 | 0 | 2
  China | 17 | 18 | 10 | 6 | 51
  Poland | 27 | 28 | 11 | 13 | 79
  Brazil | 17 | 19 | 14 | 10 | 60
  France | 0 | 1 | 0 | 1 | 2
  Serbia | 18 | 15 | 3 | 7 | 43
  Chile | 12 | 7 | 4 | 4 | 27
  Croatia | 3 | 1 | 1 | 1 | 6
  Colombia | 11 | 13 | 8 | 7 | 39
  Argentina | 21 | 23 | 13 | 16 | 73
  Romania | 11 | 6 | 3 | 4 | 24
  Hungary | 16 | 13 | 5 | 5 | 39
  Japan | 6 | 9 | 4 | 5 | 24
  Philippines | 13 | 8 | 5 | 7 | 33
  United Kingdom | 3 | 3 | 3 | 1 | 10
  Switzerland | 0 | 0 | 2 | 0 | 2
  India | 20 | 20 | 13 | 12 | 65
  Spain | 3 | 9 | 6 | 3 | 21
  Belgium | 1 | 1 | 1 | 0 | 3
  Taiwan | 8 | 10 | 5 | 7 | 30
  Italy | 2 | 0 | 1 | 1 | 4
  Mexico | 40 | 40 | 15 | 17 | 112
  South Africa | 13 | 9 | 6 | 6 | 34
  Israel | 3 | 3 | 0 | 0 | 6
  Australia | 5 | 6 | 4 | 2 | 17
  Germany | 9 | 11 | 4 | 5 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Percentage of participants with TEAEs. A treatment-emergent AE (TEAE) is defined as an event that first occurred or worsened in severity after the first dose of study treatment in Study JAIM and on or prior to the last visit date during the analysis period. The analysis period is defined as the treatment period plus up to 30 days off-drug follow-up time.
  A summary of serious and other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Week 134
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | Placebo to 2 mg Baricitinib | Placebo to 4 mg Baricitinib
Number analyzed (Participants) | 388 | 378 | 189 | 191
Percentage of Participants | 61.9 | 68.8 | 65.1 | 64.4

2. Primary Outcome: Percentage of Participants With Adverse Events of Special Interest (AESIs)
Description: Percentage of Participants with AESIs. AESI consisted of infections, positively adjudicated arterial thromboembolic events (ATE), positively adjudicated venous thromboembolic events (VTE), positively adjudicated major adverse cardiovascular events (MACE), other positively adjudicated cardiovascular events, death, anaphylactic reactions, hypersensitivity, angioedema, and malignancies.
Time Frame: Week 134
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | Placebo to 2 mg Baricitinib | Placebo to 4 mg Baricitinib
Number analyzed (Participants) | 388 | 378 | 189 | 191
Percentage of participants
  Infections | 38.4 | 42.1 | 36.5 | 35.1
  Positively adjudicated ATE | 0.3 | 0.8 | 0.5 | 0.5
  Positively adjudicated VTE | 0.3 | 1.1 | 0.5 | 0.5
  Positively adjudicated MACE | 0.3 | 0.8 | 0.5 | 0.5
  Other positively adjudicated cardiovascular events | 0.3 | 0.8 | 0 | 0.5
  Death | 0 | 1.6 | 1.1 | 0
  Anaphylactic reactions | 3.6 | 4.2 | 5.8 | 3.1
  Hypersensitivity | 3.6 | 4.2 | 5.8 | 3.1
  Angioedema | 1.3 | 0.8 | 1.6 | 0
  Malignancies | 0.5 | 0.3 | 0 | 0

3. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: Percentage of participants with SAEs. An SAE is any AE from this study that results in one of the following outcomes: Death; Initial or prolonged inpatient hospitalization; A life-threatening experience (that is, immediate risk of dying); Persistent or significant disability/incapacity; Congenital anomaly/birth defect; Important medical events that may not be immediately life-threatening or result in death or hospitalization, but may jeopardize the patient or may require intervention to prevent one of the other outcomes listed in the definition above.
  A summary of all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Week 134
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | Placebo to 2 mg Baricitinib | Placebo to 4 mg Baricitinib
Number analyzed (Participants) | 388 | 378 | 189 | 191
Percentage of Participants | 11.1 | 13.5 | 11.1 | 11.5

4. Primary Outcome: Percentage of Participants With Temporary Investigational Product Interruptions
Description: Percentage of participants with temporary investigational product interruptions.
Time Frame: Week 134
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | Placebo to 2 mg Baricitinib | Placebo to 4 mg Baricitinib
Number analyzed (Participants) | 388 | 378 | 189 | 191
Percentage of Participants | 19.1 | 24.6 | 18.5 | 23.6

5. Primary Outcome: Percentage of Participants With Permanent Investigational Product Discontinuations
Description: Percentage of participants with permanent investigational product discontinuations.
Time Frame: Week 134
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | Placebo to 2 mg Baricitinib | Placebo to 4 mg Baricitinib
Number analyzed (Participants) | 388 | 378 | 189 | 191
Percentage of Participants | 5.2 | 5.8 | 4.2 | 5.8

6. Secondary Outcome: Percentage of Participants Achieving a Systemic Lupus Erythematosus Responder Index 4 (SRI-4) Response
Description: SRI-4 response defined as 1)greater than or equal to 4-point reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) total score 2)no new British Isles Lupus Assessment Group (BILAG) A and no more than 1 new BILAG B domain score and 3)no worsening in Physician Global Assessment (PGA) of Disease Activity (worsening defined as an increase of >=0.3 from baseline on a 0-3 visual analogue scale).
  SLEDAI-2K assessment consists of 24 items with total score of 0(no symptoms) to 105 (presence of all defined symptoms) with higher scores representing increased disease activity. BILAG Index: assessing clinical signs, symptoms,or laboratory parameters related to Systemic Lupus Erythematosus (SLE),divided into 9 organ systems. For each organ system A=severe disease,B=moderate disease,C=mild stable disease,D=inactive,but previously active,E=inactive and never affected. PGA assesses disease activity on a visual analogue scale from 0 to 3 (1=mild, 2=moderate, 3=severe).
Time Frame: Week 134
Population: All randomized participants who had SLEDAI-2K score of >=4 at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | Placebo to 2 mg Baricitinib | Placebo to 4 mg Baricitinib
Number analyzed (Participants) | 388 | 379 | 129 | 131
Percentage of participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants Achieving a Lupus Low Disease Activity State (LLDAS)
Description: Percentage of participants achieving a LLDAS. The LLDAS is a composite measure designed to identify patients achieving a state of low disease activity. The LLDAS response criteria were: (1) SLEDAI-2K <=4, with no activity in major organ systems (CNS, vascular, renal, cardiorespiratory and constitutional); where "no activity" is defined as all items of SLEDAI-2K within these major organ systems equal to 0. (2) no new features of lupus disease activity compared to previous occurred visit, where the "new feature" is defined as any of the SLEDAI-2K 24 items changed from 0 to greater than 0; (3) PGA (scale 0-3), <=1; (4) current prednisolone (or equivalent) dose <=7.5 mg daily.
Time Frame: Week 48
Population: All participants who received at least one dose of study drug and had SLEDAI-2K score of >=4 at baseline. Due to early termination of the study, this population consisted of participants who completed Week 48 treatment, or discontinued treatment prior to Week 48 (but not due to study termination).
Measure: Number; unit: Percentage of participants
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | Placebo to 2 mg Baricitinib | Placebo to 4 mg Baricitinib
Number analyzed (Participants) | 289 | 261 | 98 | 100
Percentage of participants | 29.8 | 33.0 | 19.4 | 26.0

8. Secondary Outcome: Change From Baseline in Prednisone Dose
Description: Change from baseline in prednisone dose.
Time Frame: Baseline through Week 48
Population: Due to early termination of the study, this population consisted of participants who completed Week 48 treatment, or discontinued treatment prior to Week 48 (but not due to study termination). Participants having values for this outcome were included.
Measure: Least Squares Mean (Standard Error); unit: milligrams (mg)
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | Placebo to 2 mg Baricitinib | Placebo to 4 mg Baricitinib
Number analyzed (Participants) | 235 | 225 | 115 | 121
milligrams (mg) | 2.35 (0.305) | 2.27 (0.316) | 1.68 (0.426) | 1.00 (0.419)

9. Secondary Outcome: Annualized Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA)-Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) Flare Index Flare Rate
Description: The SELENA-SLEDAI tool is a cumulative and weighted index used to assess disease activity across 24 different disease descriptors in patients with lupus. A patient's SELENA-SLEDAI total score is the sum of all marked lupus related descriptors (seizure, psychosis, organic brain syndrome, visual disturbance, cranial nerve disorder, lupus headache, cerebrovascular accident, vasculitis, arthritis, myositis, urinary casts, hematuria, proteinuria, pyuria, new rash, alopecia, mucosal ulcers, pleurisy, pericarditis, low complement, increased DNA binding, fever, thrombocytopenia, leukopenia). A total score can fall between 0 and 105, with a higher score representing a more significant degree of disease activity. The annualized flare rate is calculated as the number of flares divided by the flare exposure time in days multiplied with 365.25.
Time Frame: Baseline through Week 48
Population: as for outcome 8
Measure: Number; unit: flares per year
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | Placebo to 2 mg Baricitinib | Placebo to 4 mg Baricitinib
Number analyzed (Participants) | 289 | 261 | 136 | 143
flares per year | 0.978 | 0.926 | 0.894 | 0.746

10. Secondary Outcome: Percentage of Participants With Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Total Activity Score ≥10 at Baseline With ≥50% Reduction in CLASI Total Activity Score
Description: The CLASI is a single-page tool that separately quantifies disease activity and damage. For the activity score, points are given for the presence of erythema, scale, mucous membrane lesions, recent hair loss, and inflammatory alopecia. The total score represents the sum of the individual scores and ranges from 0 to 70. Higher scores are awarded for more severe manifestations.
Time Frame: Week 48
Population: All participants with CLASI Total Activity Score >= 10 at baseline. Due to early termination of the study, this population consisted of participants who completed Week 48 treatment, or discontinued treatment prior to Week 48 (but not due to study termination).
Measure: Number; unit: Percentage of participants
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | Placebo to 2 mg Baricitinib | Placebo to 4 mg Baricitinib
Number analyzed (Participants) | 59 | 50 | 5 | 5
Percentage of participants | 55.9 | 64.0 | 60.0 | 20.0

11. Secondary Outcome: Change From Baseline in Tender Joint Count
Description: The number of tender and painful joints is determined by examination of 28 joints (14 on each side) which include: the 2 shoulders, the 2 elbows, the 2 wrists, the 10 metacarpophalangeal joints, the 2 interphalangeal joints of the thumb, the 8 proximal interphalangeal joints, and the 2 knees. The joints are assessed and classified as tender or not tender. LS mean was calculated using Mixed Model Repeated Measures (MMRM) analysis with treatment, baseline disease activity (total SLEDAI-2K <10; >=10), baseline corticosteroid dose (<10 mg/day; >=10 mg/day prednisone or equivalent), region (North America, Central/South America/Mexico, Europe, Asia and Rest of World), visit (as categorical variable), baseline value, treatment-by-visit interaction, and baseline value-by-visit interaction.
Time Frame: Baseline through Week 48
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: tender joints
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | Placebo to 2 mg Baricitinib | Placebo to 4 mg Baricitinib
Number analyzed (Participants) | 230 | 217 | 113 | 119
tender joints | -5.68 (0.281) | -5.85 (0.292) | -3.62 (0.383) | -3.73 (0.376)

12. Secondary Outcome: Change From Baseline in Swollen Joint Count
Description: The number of swollen joints is determined by examination of 28 joints (14 on each side) which include: the 2 shoulders, the 2 elbows, the 2 wrists, the 10 metacarpophalangeal joints, the 2 interphalangeal joints of the thumb, the 8 proximal interphalangeal joints, and the 2 knees. The joints are assessed and classified as swollen or not swollen. LS mean was calculated using MMRM analysis with treatment, baseline disease activity (total SLEDAI-2K <10; >=10), baseline corticosteroid dose (<10 mg/day; >=10 mg/day prednisone or equivalent), region (North America, Central/South America/Mexico, Europe, Asia and Rest of World), visit (as categorical variable), baseline value, treatment-by-visit interaction, and baseline value-by-visit interaction.
Time Frame: Baseline trough Week 48
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: swollen joints
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | Placebo to 2 mg Baricitinib | Placebo to 4 mg Baricitinib
Number analyzed (Participants) | 230 | 217 | 113 | 119
swollen joints | -4.03 (0.191) | -4.01 (0.196) | -3.19 (0.264) | -2.94 (0.257)

13. Secondary Outcome: Change From Baseline in Systemic Lupus International Collaborating Clinics/American College of Rheumatology (SLICC/ACR) Damage Index Total Score
Description: The SLICC/ACR damage index is a validated instrument to assess damage, defined as irreversible impairment, continuously persistent for 6 months (ascertained by clinical assessment), occurring since the onset of lupus, and it is based on a weighted scoring system. This index records damage occurring in participants with SLE regardless of cause, with demonstrated content, face, criterion, and discriminant validity. A score of 0 indicates no damage. Total maximum score is 47 and increasing score indicates increasing disease severity.
Time Frame: Baseline through Week 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | Placebo to 2 mg Baricitinib | Placebo to 4 mg Baricitinib
Number analyzed (Participants) | 235 | 226 | 115 | 121
Score on a scale | -0.03 (0.569) | -0.04 (0.544) | -0.04 (0.754) | -0.06 (0.505)

14. Secondary Outcome: Change From Baseline in Worst Pain Numeric Rating Scale (NRS)
Description: Change from baseline in Worst Pain NRS. It is assessed using an 11-point Numeric Rating Scale (NRS) (0-10) where 0 represents "no pain" and 10 represents "worst pain imaginable". Overall severity of a patient's pain is indicated by selecting the number that best describes the worst level of pain during the past 7 days.
Time Frame: Baseline through Week 48
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | Placebo to 2 mg Baricitinib | Placebo to 4 mg Baricitinib
Number analyzed (Participants) | 220 | 207 | 111 | 118
Score on a scale | -0.96 (0.167) | -1.23 (0.173) | -0.55 (0.222) | -0.83 (0.218)

ADVERSE EVENTS:
Time Frame: Baseline through Study Completion (Up to 134 Weeks)
Description: All participants who received at least one dose of study drug in Study JAIM and who did not discontinue from the study for the reason of Lost to Follow-up at the first post baseline visit (Safety Population). Gender specific events occurring only in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib | Placebo to 2 mg Baricitinib | Placebo to 4 mg Baricitinib
All-Cause Mortality (participants affected / at risk) | 0/388 | 6/378 | 2/189 | 0/191
Serious Adverse Events (participants affected / at risk) | 43/388 | 53/378 | 21/189 | 22/191
Other Adverse Events (participants affected / at risk) | 54/388 | 54/378 | 35/189 | 29/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 2 mg Baricitinib (N=388) | 4 mg Baricitinib (N=378) | Placebo to 2 mg Baricitinib (N=189) | Placebo to 4 mg Baricitinib (N=191)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Scleritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Immune-mediated hepatic disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acinetobacter sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 7 (7) | 3 (3) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 5 (5) | 5 (5) | 0 (0) | 3 (3)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1) | 1 (2) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 1/361 (1) | 0/356 (0) | 0/181 (0) | 0/176 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (3) | 2 (2)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Biopsy (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (6) | 1 (1) | 3 (3)
Tendon sheath disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extranodal marginal zone b-cell lymphoma (malt type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Her2 positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/361 (0) | 0/356 (0) | 1/181 (1) | 0/176 (0)
Autoimmune neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Central nervous system lupus (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/361 (0) | 1/356 (1) | 0/181 (0) | 0/176 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 2/361 (2) | 1/356 (1) | 0/181 (0) | 0/176 (0)
Endometriosis (Reproductive system and breast disorders) | 0/361 (0) | 1/356 (2) | 0/181 (0) | 0/176 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical conisation (Surgical and medical procedures) | 0/361 (0) | 0/356 (0) | 1/181 (1) | 0/176 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fasciotomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accelerated hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg Baricitinib (N=388) | 4 mg Baricitinib (N=378) | Placebo to 2 mg Baricitinib (N=189) | Placebo to 4 mg Baricitinib (N=191)
Covid-19 (Infections and infestations) | 35 (35) | 32 (33) | 21 (22) | 23 (25)
Urinary tract infection (Infections and infestations) | 20 (28) | 22 (27) | 17 (19) | 7 (8)

LIMITATIONS AND CAVEATS:
This study was terminated due to insufficient evidence to support a positive benefit: risk profile. Safety findings were consistent with previously published OLUMIANT data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT03843125/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT03843125/SAP_001.pdf